CLINICAL TRIAL: NCT03082066
Title: Assessment of Soft Tissue and Bone Diameter for Intraosseus Access in Children and Adults
Brief Title: Soft Tissue and Bone Diameter in Children and Adults for Intraosseus Access
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Collaborators: Ruth Kröss, MD EDAIC (Unknown); Glodny Bernhard, MD PD Assoc. Prof. (Unknown); Laura Trefzer, Cand med (Unknown); Sabrina Neururer, DI BSc (Unknown)
Responsible Party: Principal Investigator, Peter Paal, PD MD MBA EDAIC EDIC, MD PD MBA EDAIC EDIC, Medical University Innsbruck
Other Study IDs: AN2015-0093 348/4.17
Record Dates: First submitted 2017-02-27; First posted 2017-03-17 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Emergencies; Infusion Site Injury; Bone Infection
Keywords: bone access; intraosseus needle; resuscitation; infusion; volume therapy; emergency
MeSH Terms: conditions — Emergencies | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Younger 18 years: Newborns, infants, small child, school child, teens
  Interventions: Other: CT or MRI scan
- Adults: Even or older 18 years
  Interventions: Other: CT or MRI scan

INTERVENTIONS:
Other: CT or MRI scan — CT or MRI performed for underlying disease. CT and MRI scans used to asses bone and soft tissue diameter

SUMMARY:
Retrospective observational study: Soft tissue and bone diameters are assessed in MRI and CT scans of patients. Data is compared with recommendations of intraosseus needle producers to assess whether the information provided by the producers can be optimised. Study sites are head of humerus bone, distal femur, proximal and distal tibia in accordance with recommended intraosseus access sites.

Primary and secondary outcome parameters will be assessed at one time only, i.e. when the patient has received MRI or CT scan for the diagnostic work up of their primary disease. Data collection for a given patient in this study can be completed within one session, e.g. 5-10 minutes. No additional investigation is required for this retrospective study.

DETAILED DESCRIPTION:
Retrospective observational single centre study: Soft tissue and bone diameters are assessed in MRI and CT scans of patients. Data is compared with recommendations of intraosseus needle producers to assess whether the information provided by the producers can be optimised. Study sites are head of humerus bone, distal femur, proximal and distal tibia in accordance with recommended intraosseus access sites. Data is gathered from patients who undergo either MRI or CT scanning for any disease and where bone at the IO puncture site is accessible for measurements required for this study.

Primary and secondary outcome parameters will be assessed at one time only, i.e. when the patient has received MRI or CT scan for the diagnostic work up of their primary disease. Data collection for a given patient in this study can be completed within one session, e.g. 5-10 minutes. No additional investigation is required for this

ELIGIBILITY:
Inclusion Criteria:

* Patients 0-90 years of age with elective or emergency MRI or CT scan within a 24 months period at the university hospital Innsbruck, Austria. Patients in analgosedation, anaesthesia, and stand-by

Exclusion Criteria:

* Pathologies at recommended intraosseus puncture - and investigation- site, i.e. proximal humerus, distal femur, proximal and distal tibia

Ages: 0 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients 0-90 years of age with elective MRI or CT scan within a 24 months period at the university hospital Innsbruck, Austria. Patients in analgosedation, anaesthesia, and stand-by
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Soft tissue diameter | Retrospective single time measurement on MRI or CT scan. Measurement will last approx. 10 minutes, an will happen only once
  CT or MRI performed for underlying disease. Diameter of soft tissue at the site of recommended intraosseus bone access

SECONDARY OUTCOMES:
Bone tissue diameter | Retrospective single time measurement on MRI or CT scan.Measurement will last approx. 10 minutes, an will happen only once
  CT or MRI performed for underlying disease. Diameter of bone cortical and spongiosa at the site of recommended intraosseus bone access

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No